CLINICAL TRIAL: NCT00376324
Title: An Open-Label, Multiple-Dose Study of the Pharmacokinetics of Tigecycline in Human Bone
Brief Title: Study Evaluating the Pharmacokinetics of Tigecycline in Human Bone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-119
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
Keywords: pharmacokinetics; human bone
MeSH Terms: interventions — Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tigecycline — Each subject will receive 3 IV doses of tigecycline, as 30-minute infusions: Dose 1 = 100 mgDose 2 = 50 mgDose 3 = 50 mg The doses of tigecycline will be administered to the subjects at approximately 12-hour intervals.

SUMMARY:
Study to examine the concentration of the study drug, tigecycline, in human bone samples following the administration of multiple doses.

ELIGIBILITY:
Inclusion:

* Men and nonlactating and nonpregnant women greater than or equal to 18 years of age.
* Healthy as determined by the investigator on the basis of medical history, physical examination, vital signs, and 12-lead electrocardiogram (ECG).
* Have a high probability for compliance with and completion of the study.

Exclusion:

* Subjects with chronic osteomyelitis.
* Subjects who have known or suspected hypersensitivity to tigecycline or other tetracyclines.
* Involvement in other investigational studies of any type within 30 days before test article administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine both the bone and corresponding serum concentration of tigecycline at selected time points following adminstration. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Phoenix, Arizona, United States

REFERENCES:
- [Derived] Bhattacharya I, Gotfried MH, Ji AJ, Saunders JP, Gourley I, Diehl A, Korth-Bradley JM. Reassessment of tigecycline bone concentrations in volunteers undergoing elective orthopedic procedures. J Clin Pharmacol. 2014 Jan;54(1):70-4. doi: 10.1002/jcph.201. Epub 2013 Oct 24. PMID 24155157